CLINICAL TRIAL: NCT06917638
Title: Clinical Evaluation of Dental Implant Stability Placed in Healed Bony Sites Using Oversized Drilling Versus Conventional Drilling Protocol: A Randomized Controlled Clinical Trial
Brief Title: Dental Implant Stability Placed in Healed Bony Sites Using Oversized Drilling Versus Conventional Drilling Protocol
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ِAmr Said Ahmed el sayed el shikh, Masters student, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: https://cu.edu.eg/ar/Home
Record Dates: First submitted 2024-03-17; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Implant Complication
Keywords: implant stability

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will be randomly selected into either group using computer generated randomization using (www.randomizer.org).
  The randomized numbers will be allocated to each site in each patient and will be placed in opaque, sealed and sequentially numbered envelopes. Patients will be randomly allocated to test and control groups using the randomization schedule.
  Masking/blinding:
  * Participants will be blinded.
  * Blinding of the operator will not be applicable
  * The outcome assessor will be blinded
  * The biostatistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: Under-sized drilling group (UD) (Active Comparator): Manufacturer-recommended implant osteotomy preparation will be done according to the manufacturer guidelines with the final drill the same diameter of the implant.
  Interventions: Procedure: implant placment
- Intervention Group: oversized drilling (OD) (Active Comparator): Osteotomy preparations for the oversized drilling group will include an extra drill, which will be 0.2mm wider than the diameter of the implant.
  Interventions: Procedure: implant placment

INTERVENTIONS:
Procedure: implant placment — * Crestal incision followed by full thickness mucoperiosteal flap elevation.
  * Drilling of the implant according to the manufacturer's instructions to reach the final drill corresponding to the implant size.
  * Allocation concealment will be broken at this point to assign the patient into one of two groups:
  Control Group: osteotomy preparation the same diameter of the implant. Intervention: oversized drilling:Osteotomy preparations will include an extra drill,(0.2mm) wider than the diameter of the implant.
  * A smart peg will then be attached to the implant, to measure its stability using Ostell and three readings will be recorded:occlusal buccal and lingual reading.
  * A healing collar will then be place over the implant, then simple intrerupted suture
  * A standardized digital periapical radiograph will be taken using a radiographic holder and a custom-made radiographic stent to determine the initial crestal bone level.

SUMMARY:
The goal of this [type of study: clinical trial] is to [investigate the influence of Oversized Drilling Versus Traditional for implant Stability and Crestal Bone Loss.] in [ Healthy Patient aged between 20 and 60 years with one missing tooth in the posterior mandible with sufficient bone dimensions].

The main question[s] it aims to answer are:

the influence of oversized drilling versus traditional drilling in the mandibular arch, in terms of implant stability and crestal bone levels. The effects of oversized protocol have not been fully explored on the more compact mandibular bone.

Participants will Control Group: Under-sized drilling group (UD):

Manufacturer-recommended implant osteotomy preparation will be done according to the manufacturer guidelines with the final drill the same diameter of the implant. Intervention Group: oversized drilling (OD) Osteotomy preparations for the oversized drilling group will include an extra drill, which will be 0.2mm wider than the diameter of the implant.

* Once the osteotomy is ready, the appropriate implant will be placed manually at first and then progressed using a ratchet.
* After the implant is correctly placed, a smart peg will be attached to the implant via hand screwing, to measure its stability using Ostell and four readings will be recorded: a mesial, distal, buccal and lingual reading.
* The smart peg will then be removed and will be replaced with a healing collar above the gingival margin.
* The flap will then be sutured back to its original position around the healing collar with an interrupted suture.
* A standardized digital periapical radiograph will be taken using a radiographic holder and a custom-made radiographic stent to determine the initial crestal bone level.

DETAILED DESCRIPTION:
• Pre-operative evaluation

Clinical examination:

* Evaluation of the general condition of the oral cavity of the patients will be performed to make sure it will comply with the criteria required to be enrolled in the study in terms of oral hygiene, pathological conditions, and inter-arch space.
* When the patients meet the clinical selection criteria, radiographic examination will follow.

Radiographic examination:

* A pre-operative periapical x-ray will be performed for each of the patients who met the clinical selection criteria to increase chances of eligibility prior to a pre-operative Cone Beam Computed Tomography (CBCT). This will be done to avoid unnecessary extra expenses of a CBCT and unnecessary radiation exposure.
* A pre-operative CBCT will be performed for each of the patients who met the clinical and primary radiographic selection criteria to ensure eligibility prior to the surgery.

From the obtained CBCT, the bone height, width and density will be determined.

* Once the patients passes both the clinical and radiographic selection criteria, they will be enrolled by the investigator into the study.
* The enrolled patients will then be provided with a full explanation of the aim and benefits of the study in plain language, then, given the chance to have an informed discussion with the investigator.
* Once the patients approve the intervention and agree to comply with the study guidelines, they will sign a written informed consent form translated in Arabic.

Patient preparation:

* The enrolled participants will be prepared 2 weeks prior to the surgery. This will include professional scaling, oral hygiene instructions and treatment of any caries or defective fillings present around the surgical site.
* Diagnostic impressions will be taken using alginate impression material during the preparation phase.
* After the cast is poured out, a radiographic stent will be created at the area of interest using cold cure acrylic material. This will be done by the aid of an x-ray holder consisting of an acrylic customized bite block, a metallic indicator arm and a radiographic rim. The aim of this step is to standardize the position of the digital xray for each site in order to ensure reproducibility between follow ups when measuring crestal bone loss.

  - Surgical procedure:
* After local anaesthesia, a crestal incision will be performed at the site using a 15c blade followed by full thickness mucoperiosteal flap elevation to expose the underlying bone. A periodontal probe will then be used to help locate the correct point of drilling. This will be done by leaving a margin(1mm) between the buccal plate and the osteotomy, a margin(1mm) between the lingual plate and the osteotomy, A margin(1.5mm) between the neighboring tooth and the osteotomy.
* A round bur will used to mark the point of drilling located by the periodontal probe.
* The drilling (1200 rpm) will then performed under copious irrigation with normal saline sequentially according to the manufacturer's instructions to reach the final drill corresponding to the implant size.
* Allocation concealment will be broken at this point to assign the patient into one of two groups:

Control Group: Under-sized drilling group (UD):

Manufacturer-recommended implant osteotomy preparation will be done according to the manufacturer guidelines with the final drill the same diameter of the implant. Intervention Group: oversized drilling (OD) Osteotomy preparations for the oversized drilling group will include an extra drill, which will be 0.2mm wider than the diameter of the implant.

* Once the osteotomy is ready, the appropriate implant will be placed manually at first and then progressed using a ratchet.
* After the implant is correctly placed, a smart peg will be attached to the implant via hand screwing, to measure its stability using Ostell and four readings will be recorded: a mesial, distal, buccal and lingual reading.
* The smart peg will then be removed and will be replaced with a healing collar above the gingival margin.
* The flap will then be sutured back to its original position around the healing collar with an interrupted suture.
* A standardized digital periapical radiograph will be taken using a radiographic holder and a custom-made radiographic stent to determine the initial crestal bone level.

Postoperative instructions and follow up:

The patient will be instructed to take:

- Antibiotics (Amoxicillin 1g twice daily for 5 days) to prevent any chance of infection.

(Eugenio Romeo et al, 2014).

* Anti-inflammatory drugs (NSAIDS; Ibuprofen 600mg three times daily for 5 days) to avoid any chance of oedema or pain or swelling (Francesco pieri et al, 2012).
* Antiseptic mouth rinse (0.12% Chlorhexidine oral rinse will be prescribed for 60 seconds two times a day for 14 days. (Jun Yu et al, 2015)

The patient will be instructed to:

* Apply an ice pack to the treated area for the first 24 hours. (Francesco pieri et al, 2012).
* Avoid any brushing or trauma to the surgical site for one week. (Francesco pieri et al, 2012). The patient will be instructed to come in for weekly follow ups over the course of the following 3 months after implant placement for recording Ostell readings. After 6 months following the implant placement, (Paolantoni et al. 2013) healing collar will be removed, and impressions (indirect, open or closed tray technique) will be taken to fabricate the final crowns followed by crown placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a single missing tooth in the posterior region of the mandibular arch.
* Bone dimensions buccolingual (not less than 6mm) and apicocoronal (not less than 10mm)
* Patients with healthy systemic condition. (Brightman. 1994)
* Patients aged from 20 to 60 years old.
* Good oral hygiene. (Wiesner et al. 2010)
* Accepts 6 months follow-up period (cooperative patients)

Exclusion Criteria:

* Patients with signs of acute infection related to the area of interest.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as parafunctional habits or alcoholism (Lobbezoo et al. 2006).
* Smokers (Bruno Ramos Chrcanovic et al. 2015) (25).
* Pregnant women
* Patients on medication that may interfere with healing (corticosteroids, bisphosphonate, Chemo/radio therapy).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
Implant stability quotient (ISQ) | 1 week, 2 weeks, 3 weeks, 4 weeks, 6 weeks, 8 weeks, and 12 weeks postoperatively.
  resonance frequency analysis

SECONDARY OUTCOMES:
• crestal bone levels (day of the surgery (baseline), at 3 and 6 months postoperatively) • pain • swelling • satisfaction • implant survival | (day of the surgery (baseline), at 3 and 6 months postoperatively)
  parallel technique periapical radiography
  VAS Categorical scale Questionnaire Categorical scale

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seleem A, Tawfik OK, El-Nahass H. Evaluation of Oversized Drilling on Implant Survival and Stability Versus Traditional Drilling Technique: A Randomized Clinical Trial. Int J Oral Maxillofac Implants. 2021 Jul-Aug;36(4):771-778. doi: 10.11607/jomi.8777. PMID 34411219
- See also: Oversized implants — https://pubmed.ncbi.nlm.nih.gov/34411219/